CLINICAL TRIAL: NCT04877340
Title: Prospective Randomized Study Comparing the 25-gauge Franseen Needle and the 25-gauge Standard Needle for EUS-guided Fine-needle Sampling of Solid Pancreatic Lesions Without Rapid on Site Evaluation
Brief Title: Comparation Between Needles for EUS-guided Sampling of Solid Pancreatic Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 26962419.3.0000.0065
Record Dates: First submitted 2021-04-20; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Pancreatic Neoplasms
Keywords: accuracy; pancreatic cancer; endoscopic ultrasound-guided
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard FNA 22G needle (Other): The pancreatic mass will be puncture, for expert endoscopist, with a standard FNA 22G needle
  Interventions: Device: needle punction
- Franseen 22G needle (Experimental): The pancreatic mass will be puncture, for expert endoscopist, with a FNB 22G needle. The sequence of the use of needles will be randomized.
  Interventions: Device: needle punction

INTERVENTIONS:
Device: needle punction — EUS-guided sampling of pancreatic solid lesions obtained with the 22-gauge

SUMMARY:
This is a randomized study in order to compare the diagnostic yield (primary outcome) of EUS-guided sampling of pancreatic solid lesions obtained with the 25-gauge Franseen and the 25-gauge standard needle in patients undergoing EUS-guided sampling of pancreatic solid masses without ROSE. Secondary outcomes are the number of extra passes with each needle required to reach adequate core, possibility to perform immunohistochemistry and the adverse event rate.

DETAILED DESCRIPTION:
This is a randomized trial conducted at a unique center. The aim of this study is to compare the diagnostic yield (primary outcome) of EUS-guided sampling of pancreatic solid lesions obtained with the 25-gauge Franseen and the 25-gauge standard needle in patients undergoing EUS-guided sampling of pancreatic solid masses without ROSE. Secondary outcomes are the number of extra passes with each needle required to reach adequate core, possibility to perform immunohistochemistry and the adverse event rate.

Patients with a suspected solid pancreatic lesion larger than 15 mm, identified by CT or MRI and referred to EUS-guided sampling will be eligible for inclusion. Patients will be excluded in case of cystic lesion, or the lesion was not detected in EUS, or if the coagulation parameters are abnormal (INR> 2, platelet count < 50,000). The pancreatic mass will be puncture, for expert endoscopist, firstly with a needle according to randomization, followed by another one. Will be make a touch print with the specimen obtained with the needles and, subsequently, all the specimen will be put in formaldehyde solution for cell-block analysis.

Diagnostic yield of cell block will be defined as enough histologic tissue core containing pancreatic parenchyma or tumor with dysplastic cells enough for the correct tissue diagnosis. In the presence of malignant tissue in core specimens, it will be calculated the proportion of the area positive for malignancy compared to the total area of the core and then the each needle yield will be defined.

ELIGIBILITY:
Inclusion Criteria:

- solid pancreatic lesion larger than 15 mm

Exclusion Criteria:

* pancreatic cystic lesion
* lesion not detected in EUS
* abnormal coagulation parameters (INR> 2, platelet count < 50,000)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11-26 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Compare the diagnostic yield | 2 years
  compare the diagnostic yield between two EUS needles

SECONDARY OUTCOMES:
extra passes with each needle | 2 years
  number of extra passes with each needle required to reach adequate core, possibility to perform immunohistochemistry
perform immunohistochemistry | 2 years
  need to perform immunohistochemistry to reach the result
adverse event rate | 2 years
  to assess the adverse event rate

CONTACTS AND LOCATIONS:
Overall Officials: FAUZE MALUF-FILHO, PHD, Principal Investigator — ICESP/FMUSP
Locations (1):
- ICESP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madhoun MF, Wani SB, Rastogi A, Early D, Gaddam S, Tierney WM, Maple JT. The diagnostic accuracy of 22-gauge and 25-gauge needles in endoscopic ultrasound-guided fine needle aspiration of solid pancreatic lesions: a meta-analysis. Endoscopy. 2013;45(2):86-92. doi: 10.1055/s-0032-1325992. Epub 2013 Jan 10. PMID 23307148
- [Background] Puri R, Vilmann P, Saftoiu A, Skov BG, Linnemann D, Hassan H, Garcia ES, Gorunescu F. Randomized controlled trial of endoscopic ultrasound-guided fine-needle sampling with or without suction for better cytological diagnosis. Scand J Gastroenterol. 2009;44(4):499-504. doi: 10.1080/00365520802647392. PMID 19117242
- [Background] Wani S, Early D, Kunkel J, Leathersich A, Hovis CE, Hollander TG, Kohlmeier C, Zelenka C, Azar R, Edmundowicz S, Collins B, Liu J, Hall M, Mullady D. Diagnostic yield of malignancy during EUS-guided FNA of solid lesions with and without a stylet: a prospective, single blind, randomized, controlled trial. Gastrointest Endosc. 2012 Aug;76(2):328-35. doi: 10.1016/j.gie.2012.03.1395. Epub 2012 Jun 12. PMID 22695205
- [Background] Itoi T, Sofuni A, Itokawa F, Irisawa A, Khor CJ, Rerknimitr R. Current status of diagnostic endoscopic ultrasonography in the evaluation of pancreatic mass lesions. Dig Endosc. 2011 May;23 Suppl 1:17-21. doi: 10.1111/j.1443-1661.2011.01132.x. PMID 21535194
- [Background] Levy MJ. Endoscopic ultrasound-guided trucut biopsy of the pancreas: prospects and problems. Pancreatology. 2007;7(2-3):163-6. doi: 10.1159/000104240. Epub 2007 Jun 21. PMID 17592229
- [Background] Fabbri C, Polifemo AM, Luigiano C, Cennamo V, Baccarini P, Collina G, Fornelli A, Macchia S, Zanini N, Jovine E, Fiscaletti M, Alibrandi A, D'Imperio N. Endoscopic ultrasound-guided fine needle aspiration with 22- and 25-gauge needles in solid pancreatic masses: a prospective comparative study with randomisation of needle sequence. Dig Liver Dis. 2011 Aug;43(8):647-52. doi: 10.1016/j.dld.2011.04.005. Epub 2011 May 17. PMID 21592873
- [Background] Wang Y, Chen Q, Wang J, Wu X, Duan Y, Yin P, Guo Q, Hou W, Cheng B. Comparison of modified wet suction technique and dry suction technique in endoscopic ultrasound-guided fine-needle aspiration (EUS-FNA) for solid lesions: study protocol for a randomized controlled trial. Trials. 2018 Jan 17;19(1):45. doi: 10.1186/s13063-017-2380-y. PMID 29343303
- [Background] Kim HJ, Jung YS, Park JH, Park DI, Cho YK, Sohn CI, Jeon WK, Kim BI, Choi KY, Ryu S. Endosonographer's macroscopic evaluation of EUS-FNAB specimens after interactive cytopathologic training: a single-center prospective validation cohort study. Surg Endosc. 2016 Oct;30(10):4184-92. doi: 10.1007/s00464-015-4727-3. Epub 2016 Jan 7. PMID 26743106
- [Background] Sadaf S, Loya A, Akhtar N, Yusuf MA. Role of endoscopic ultrasound-guided-fine needle aspiration biopsy in the diagnosis of lymphoma of the pancreas: A clinicopathological study of nine cases. Cytopathology. 2017 Dec;28(6):536-541. doi: 10.1111/cyt.12442. Epub 2017 Jul 24. PMID 28737285
- [Background] Mohanty SK, Pradhan D, Sharma S, Sharma A, Patnaik N, Feuerman M, Bonasara R, Boyd A, Friedel D, Stavropoulos S, Gupta M. Endoscopic ultrasound guided fine-needle aspiration: What variables influence diagnostic yield? Diagn Cytopathol. 2018 Apr;46(4):293-298. doi: 10.1002/dc.23883. Epub 2017 Dec 27. PMID 29280329
- [Result] Vilmann P, Jacobsen GK, Henriksen FW, Hancke S. Endoscopic ultrasonography with guided fine needle aspiration biopsy in pancreatic disease. Gastrointest Endosc. 1992 Mar-Apr;38(2):172-3. doi: 10.1016/s0016-5107(92)70385-x. No abstract available. PMID 1568614
- [Result] Iglesias-Garcia J, Dominguez-Munoz JE, Abdulkader I, Larino-Noia J, Eugenyeva E, Lozano-Leon A, Forteza-Vila J. Influence of on-site cytopathology evaluation on the diagnostic accuracy of endoscopic ultrasound-guided fine needle aspiration (EUS-FNA) of solid pancreatic masses. Am J Gastroenterol. 2011 Sep;106(9):1705-10. doi: 10.1038/ajg.2011.119. Epub 2011 Apr 12. PMID 21483464
- [Result] Iglesias-Garcia J, Poley JW, Larghi A, Giovannini M, Petrone MC, Abdulkader I, Monges G, Costamagna G, Arcidiacono P, Biermann K, Rindi G, Bories E, Dogloni C, Bruno M, Dominguez-Munoz JE. Feasibility and yield of a new EUS histology needle: results from a multicenter, pooled, cohort study. Gastrointest Endosc. 2011 Jun;73(6):1189-96. doi: 10.1016/j.gie.2011.01.053. Epub 2011 Mar 21. PMID 21420083
- [Result] Bang JY, Hebert-Magee S, Hasan MK, Navaneethan U, Hawes R, Varadarajulu S. Endoscopic ultrasonography-guided biopsy using a Franseen needle design: Initial assessment. Dig Endosc. 2017 May;29(3):338-346. doi: 10.1111/den.12769. Epub 2016 Dec 20. PMID 27878861